CLINICAL TRIAL: NCT04284215
Title: Department of Oncology, Affiliated Hospital of Guizhou Medical University
Brief Title: Efficacy and Safety of Albumin Paclitaxel Combined With Cisplatin Chemoradiotherapy for Non-resectable Stage III NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guizhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GuizhouMu
Record Dates: First submitted 2019-09-14; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2019-07

CONDITIONS: Efficacy and Safety
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin paclitaxel (Experimental): Albumin paclitaxel 40mg/m2/week was injected into normal saline at the same time as radiotherapy, once a week. Cisplatin 75 mg/m2 was given intravenously for 2-3 days , carboplatin 300 mg/m2 and 2 days. (Because toxicity and heart problems can replace DDP)] Repeat every cycle (21-28 days/cycle, minimum 2 cycles).
  Three-dimensional radiotherapy:
  intensity-modulated radiotherapy (IMRT) or rotational intensity-modulated radiation therapy (VMAT) segmented dose: primary focus and mediastinal metastatic lymph nodes; segmented mode: continuous accelerated hypersegmentation; Dose: DTGTV: > 60 Gy
  Interventions: Drug: Albumin paclitaxel combined with cisplatin
- Paclitaxel (Active Comparator): Paclitaxel 175 mg/m2 was injected into saline solution on the first day. Cisplatin 75 mg/m2 was given intravenously for 2-3 days , carboplatin 300 mg/m2 and on the second day. (Because toxicity and heart problems can replace DDP)]Repeated every cycle (21-28 days/cycle, minimum 2 cycles).
  Three-dimensional radiotherapy:
  intensity-modulated radiotherapy (IMRT) or rotational intensity-modulated radiation therapy (VMAT) segmented dose: primary focus and mediastinal metastatic lymph nodes; segmented mode: continuous accelerated hypersegmentation; Dose: DTGTV: > 60 Gy
  Interventions: Drug: Albumin paclitaxel combined with cisplatin

INTERVENTIONS:
Drug: Albumin paclitaxel combined with cisplatin — Non-resectable stage III non-small cell lung cancer is recommended for concurrent chemoradiotherapy. Paclitaxel and platinum are commonly used in chemotherapy regimens. The aim of this study was to investigate whether paclitaxel albumin combined with cisplatin combined with three-dimensional primary radiotherapy could improve short-term efficacy, local progression-free survival, and reduce treatment-related toxicity. To determine whether paclitaxel albumin combined with cisplatin regimen chemotherapy can be used as a first-line treatment for stage III non-small cell lung cancer with concurrent primary thoracic radiotherapy.
  Other Names: Albumin paclitaxel

SUMMARY:
Non-resectable stage III non-small cell lung cancer is recommended for concurrent chemoradiotherapy. Paclitaxel and platinum are commonly used in chemotherapy regimens. The aim of this study was to investigate whether paclitaxel albumin combined with cisplatin combined with three-dimensional primary radiotherapy could improve short-term efficacy, local progression-free survival, and reduce treatment-related toxicity. To determine whether paclitaxel albumin combined with cisplatin regimen can be used as a first-line treatment for stage III non-small cell lung cancer with concurrent primary thoracic radiotherapy

DETAILED DESCRIPTION:
Control group: Paclitaxel 175 mg/m2 was injected into saline solution on the first day. Cisplatin 75 mg/m2 was given intravenously for 2-3 days (2-4 days), carboplatin 300 mg/m2 and 2 days. (Because toxicity and heart problems can replace DDP)]Repeated every 3-4 weeks for 4 consecutive cycles (21-28 days/cycle, minimum 2 cycles). In the experimental group, albumin paclitaxel 40 mg/m2/week was injected into saline at the same time as radiotherapy, once a week. Cisplatin 75 mg/m2 was given intravenously for 2-3 days (2-4 days), carboplatin 300 mg/m2 and 2 days. (Because toxicity and heart problems can replace DDP)] Repeat every 3-4 weeks for 4 consecutive cycles (21-28 days/cycle, minimum 2 cycles). Three-dimensional radiotherapy: intensity-modulated radiotherapy (IMRT) or rotational intensity-modulated radiation therapy (VMAT) segmented dose: primary focus and mediastinal metastatic lymph nodes; segmented mode: continuous accelerated hypersegmentation Dose: DTGTV: > 60Gy treatment sequence: Chemotherapy started within one week after completion of pre-treatment evaluation. Radiotherapy for primary thoracic tumors was performed simultaneously on the first day of chemotherapy. Chemotherapy effectiveness was evaluated by radiological examination within one week after the completion of the second cycle of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NSCLC confirmed by pathology or cytology; clinical stage III [AJCC 8th Edition stage];
* Informed consent signed before treatment (radiotherapy, chemotherapy);
* no contraindication of radiotherapy and chemotherapy; .IMRT or VMAT technology is required to achieve the prescription dose of primary tumor (DTGTV): > 60Gy, normal lung in the design of radiotherapy plan.
* (Total Lung Volume minus GTV Volume) V20 < 32% were randomly enrolled in the study. [Planning Assessment: Prescription dose includes 100% GTV, 90% .prescription dose includes 98%~100% PTV] [Age 18-80 years old, body condition score ECOG0-2 or KPS (>70) ];
* [Subjects had no major organ dysfunction, blood routine, lung, liver and kidney. With normal function and cardiac function, laboratory tests must meet the following requirements: leukocyte (>4.0 *109/L), neutrophil (>2.0 *109/L), platelet (>100 *109/L) and hemoglobin (>100 g/L). Liver function: normal range. Renal function: normal range .Lung function: FEV1 > 50%, mild to moderate lung function impairment. _Patients have good compliance with the treatment and follow-up.

Exclusion Criteria:

* Pathological types, stages and survival status of patients who did not meet the criteria for enrollment
* Patients with uncontrollable hypertension, diabetes mellitus, unstable angina, history of myocardial infarction or symptomatic congestive heart failure or uncontrollable arrhythmia in the past 12 months; .Clinically diagnosed valvular disease; active period of bacterial, fungal or viral infections; mental disorders; and severe heart failure.
* Pulmonary impairment; Pregnancy and lactation patients;
* Patients with a history of active malignancies other than small cell lung cancer before admission;
* Patients with non-melanoma skin basal cell carcinoma, cervical cancer in situ, and cured early prostate cancer except; .Allergic constitution and known or suspected drug allergy in any study. .Patients without alternative drugs, patients with poor compliance, and researchers do not consider it appropriate to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 2 years
  Efficacy of Concurrent chemoradiotherapy

SECONDARY OUTCOMES:
Side effection | 2 years
  bone marrow suppression, hepatic and renal toxicity, cardiac toxicity, radiation pneumonia and other toxic and side effects caused by treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bing Lu, Bachelor, Principal Investigator — Affiliated Hospital of Guizhou Medical University
Locations (1):
- Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No